CLINICAL TRIAL: NCT04485923
Title: Accuracy of Body Temperature Measurements Using the Esophageal Temperature Probe Inserted Through the Gastric Lumen of Supraglottic Airway Device
Status: Completed | Type: Observational
Sponsor: Sojin Shin (Other)
Responsible Party: Sponsor-Investigator, Sojin Shin, fellow, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: SGA_temp_adult
Record Dates: First submitted 2020-07-17; First posted 2020-07-24 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Core Temperature
Keywords: core temperature, tympanic membrane, esophageal temperature, temporal artery temperature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In general, 50-90% of patients undergoing surgery under general anesthesia are known to develop hypothermia during surgery. Due to hypothermia during surgery, the patient may cause coagulation disorders, wound infections, increased ventricular tachycardia, prolonged anesthesia drug effects, and electrification, resulting in delayed recovery after surgery, extended recovery room exit, and extended hospital stay. Therefore, unless intentional hypothermia is needed, active body temperature management during surgery is necessary.

Pulmonary artery, distal esophagus, tympanic membrane, nasopharynx, oral cavity, axillary cavity, rectum, and bladder can be measured. The most accurate method for measuring deep body temperature in general anesthesia is esophageal body temperature, nasopharyngeal body temperature, It is known as tympanic body temperature. 3,4 However, the tympanic body temperature has the disadvantage that it cannot be continuously measured. Considering these points, esophageal thermometers that can be continuously measured in patients with general anesthesia and have few side effects are commonly used. The esophageal thermometer is usually inserted through the oral cavity. When the supraglottic airway device is inserted, the space in the oral cavity is filled with the supraglottic airway device, making it difficult to mount the esophageal thermometer. However, most second-generation supraglottic airway devices have gastric lumens, and gastric lumens are connected to the esophagus, allowing esophageal thermometers to be mounted through this space. Since the esophageal temperature probe is inserted in all general anesthesia patients using the supraglottic airway device in this application, the body temperature measured by the temporal artery at the same time is how accurate the body temperature measured at this time is as a reference value using the tympanic membrane. I would like to analyze the transient comparison. We will also analyze whether the esophageal thermometer mounted through the gastric lumen of the supraglottic airway device reflects the rapidly decreasing body temperature change when the pneumatic tourniquet is decompressed.

DETAILED DESCRIPTION:
Basic anesthesia management is the same as for patients undergoing general anesthesia using all supraglottic airway devices.

Fasting from midnight the day before surgery, and when the patient enters the operating room, a blood pressure monitor, electrocardiogram, pulse saturator is mounted, and baseline blood pressure, oxygen saturation, and heart rate are recorded. As an anesthesia-inducing facial mask, it provides 100% of 4-6L/min of oxygen. Propofol is administered at 2 mg/kg, and after the patient's self-breathing is lost, 5% sevoflurane is supplied for 3 minutes to deepen the depth of anesthesia. After inserting the appropriate size of supraglottic airway (i-gel) according to the patient's weight, the esophageal temperature probe is inserted through the gastric lumen to the end of the supraglottic airway device i-gel. After 10 minutes, when the body temperature measurement measured in the esophagus stabilizes, the body temperature is measured at the tympanic membrane and temporal artery at 10-minute intervals. For the objectivity of body temperature measurement, the same operator performs it, and the left and right sides of the tympanic membrane can be measured differently, so both sides are measured and averaged. After Tourniquet deflation, body temperature is measured and recorded every 10 minutes from 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adults 19 to 80 Patients with ASA PS 1-3 Among patients undergoing knee surgery using tourniquet for more than 1 hour, patients undergoing general anesthesia using the Supraglottic airway device

Exclusion Criteria:

* Patients who refuse to participate in the study Patients with esophageal tumors or varicose veins Patients who are inserted through the esophagus during surgery Patients with ear inflammation Patients who have been deemed unsuitable for participation by the medical staff for other reasons

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among patients undergoing knee surgery using tourniquet for more than 1 hour, patients undergoing general anesthesia using the Supraglottic airway device
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-07-08 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
esophageal temperature | 10min
  'c

CONTACTS AND LOCATIONS:
Overall Officials: wonwook ko, professor, Study Chair — Asan Medical Center
Locations (1):
- asanMC, Seoul, Song-pa, South Korea

IPD SHARING:
Plan to Share IPD: Undecided